CLINICAL TRIAL: NCT03542175
Title: A Phase I Study of Rucaparib Administered Concurrently With Postoperative Radiotherapy in Patients With Triple Negative Breast Cancer With an Incomplete Pathologic Response Following Neoadjuvant Chemotherapy
Brief Title: A Study of Rucaparib Administered With Radiation in Patients With Triple Negative Breast Cancer With an Incomplete Response Following Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Clovis Oncology, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-002; P50CA247749 (NIH)
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Rucaparib; Radiotherapy; Triple Negative Breast Cancer; 18-002
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — rucaparib; Radiotherapy

STUDY DESIGN:
Intervention Model Description: This is a single-arm Phase I study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rucaparib Administered With Radiation (Experimental): one dose level (200 mg BID, 200 mg QD, 300 mg BID, 300 mg QD or 400 mg BID) concurrently with a 6-week course of radiotherapy and 4 additional weeks of maintenance rucaparib at the same dose level.
  Radiotherapy will consist of 50 Gy in 2 Gy per fraction to the breast or chest wall with or without regional nodes plus a 10 Gy boost to the lumpectomy cavity, to a total dose of 60 Gy. A 10 Gy boost to the post-mastectomy scar is allowed at the discretion of the treating physician.
  Interventions: Drug: Rucaparib; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Rucaparib — one dose level (200 mg BID, 200 mg QD, 300 mg BID, 300 mg QD or 400 mg BID) concurrently with a 6-week course of radiotherapy and 4 additional weeks of maintenance rucaparib at the same dose level.
Radiation: Radiotherapy — 50 Gy in 2 Gy per fraction to the breast or chest wall with or without regional nodes plus a 10 Gy boost to the lumpectomy cavity, to a total dose of 60 Gy. A 10 Gy boost to the post-mastectomy scar is allowed at the discretion of the treating physician.

SUMMARY:
The purpose of this study is to test the safety of a study drug called Rucaparib, administered in combination with the type of radiation therapy that is usually given to women with your form of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female, ≥ 18 years of age.
* Non-metastatic, histologically or cytologically-confirmed TNBC (defined as ER <1%, PR <1%, her-2-neu 0-1+ by IHC or FISH-negative or as per MD discretion), with evidence of residual disease in the breast or lymph nodes after neoadjuvant chemotherapy, at the time of definitive surgical treatment.
* Non-metastatic, histologically or cytologically-confirmed hormone-receptor positive, Her2/neu negative breast cancer (defined as ER >1% or PR >1% AND Her-2/neu 0-1+ by IHC or FISH-negative, or as per MD discretion), with evidence of residual grade 3 invasive breast cancer AND either 1) >5 cm of residual disease in the breast OR 2) ≥ 4 axillary LNs in the axilla after neoadjuvant chemotherapy, at the time of definitive surgical treatment.
* Definitive surgical treatment with breast-conserving surgery or mastectomy and axillary lymph node evaluation.
* At least 6-month life expectancy, ECOG Performance status < 2.
* Willingness to discontinue any cytotoxic chemotherapeutic agents, and biologic therapy at least 2 weeks prior to the start of RT.
* Adequate organ function (assessed within 30 days prior to initiation of protocol treatment, unless otherwise indicated) as follows:

Hematology

* Absolute Neutrophil Count (ANC) ≥1500/mm^3
* Platelet Count ≥100,000/mm^3
* Hemoglobin ≥9.0 g/dL (after transfusion if required) Renal Function
* Creatinine Serum ≤ 1.5 mg/dL or Creatinine Clearance ≥ 45 mL/min^a Hepatic Function
* Bilirubin ≤ 1.5 mg/dL
* Aspartate Aminotransferase (AST) ≤ 2.5 x ULN^b
* Alanine Aminotransferase (ALT) ≤ 2.5 x ULN ULN = upper normal limit of institution's normal range

  1. If calculated creatinine clearance is < 45mL/min, a 24-hour urine collection for creatinine clearance may be performed
  2. Subjects with documented Gilbert's disease may have bilirubin up to 2.5 mg/dL

     * Negative serum pregnancy test within 14 days prior to study treatment if a woman has child-bearing potential. Subjects of child bearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
     * Ability to swallow and retain oral medications.
     * Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
     * Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the duration of study participation. Should a woman become pregnant while participating on study, she should inform the treating physician immediately.

Exclusion Criteria:

* Gross residual tumor on imaging or positive margins after breast conserving surgery that are un-excised, as radiation dose in the study will be limited to 60 Gy.
* Complete pathologic response to NAC.
* Receipt of PARP inhibitor prior to RT.
* Pregnant or expecting to conceive within the projected duration of the trial, starting with screening visit through 180 days after the last dose of trial treatment.
* Prior history of radiation therapy to the ipsilateral breast and/or regional nodes is not allowed (prior RT to other sites is permitted).
* Patients with breast augmentation implants are excluded.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rucaparib.
* Concomitant anti-neoplastic treatment is not allowed during protocol treatment and should be completed at least 2 weeks prior to commencement of protocol treatment, with resolution of associated acute toxicities. Bisphosphonates are permitted without restriction even during protocol treatment. Maintenance pembrolizumab is permitted during the protocol treatment.
* Significant comorbidity: Patients with clinically significant and uncontrolled major disease or disorder that could exacerbate potential toxicities, confound safety assessments, require excluded therapy for management, or limit study compliance.
* Ongoing therapy with other investigational agents. Patients may not be receiving any other investigational agents.
* Unresolved toxicity from other agents. Patients with unresolved CTCAE v4.03 Grade 3 or greater toxicity from prior administration of another investigational drug and/or anti-cancer treatment are not eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 31 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2025-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atif Khan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Norwalk Hospital, Norwalk, Connecticut
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Rucaparib 200 mg BID; Rucaparib 200 mg QD; Rucaparib 300 mg BID; Rucaparib 300 mg QD; Rucaparib 400 mg BID: Treatment will consist of rucaparib at one dose level (200 mg BID, 200 mg QD, 300 mg BID, 300 mg QD or 400 mg BID) concurrently with a 6-week course of radiotherapy and 4 additional weeks of maintenance rucaparib at the same dose level.
  Radiotherapy will consist of 50 Gy in 2 Gy per fraction to the breast or chest wall with or without regional nodes plus a 10 Gy boost to the lumpectomy cavity, to a total dose of 60 Gy. A 10 Gy boost to the post-mastectomy scar is allowed at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Rucaparib 200 mg BID | Rucaparib 200 mg QD | Rucaparib 300 mg BID | Rucaparib 300 mg QD | Rucaparib 400 mg BID
Started | 2 | 6 | 5 | 16 | 2
Completed | 2 | 6 | 5 | 16 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rucaparib 200 mg BID | Rucaparib 200 mg QD | Rucaparib 300 mg BID | Rucaparib 300 mg QD | Rucaparib 400 mg BID | Total
Number analyzed (Participants) | 2 | 6 | 5 | 16 | 2 | 31
Age, Continuous [Median (Full Range); unit: years] | 54 [33 to 75] | 54 [38 to 70] | 48 [41 to 60] | 50 [31 to 66] | 50 [36 to 59] | 50 [31 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 5 | 16 | 2 | 31
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 2 | 3 | 5 | 13 | 2 | 25
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 3 | 0 | 3
  White | 2 | 4 | 3 | 11 | 0 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 6 | 5 | 16 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities
Description: Number of Dose Limiting Toxicities encountered at each dose level. The trial will be monitored using TITE-CRM. Assuming a model for the time to occurrence of toxic response as a function of dose, the method allows information from all enrolled patients to be used when allocating a new patient to a dose level.
Time Frame: 1 year
Measure: Number; unit: Dose limiting toxicities
Arm/Group | Rucaparib 200 mg BID | Rucaparib 200 mg QD | Rucaparib 300 mg BID | Rucaparib 300 mg QD | Rucaparib 400 mg BID
Number analyzed (Participants) | 2 | 6 | 5 | 16 | 2
Dose limiting toxicities | 1 | 0 | 3 | 3 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rucaparib 200 mg BID | Rucaparib 200 mg QD | Rucaparib 300 mg BID | Rucaparib 300 mg QD | Rucaparib 400 mg BID
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/6 | 0/5 | 4/16 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/6 | 0/5 | 1/16 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 6/6 | 5/5 | 16/16 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib 200 mg BID (N=2) | Rucaparib 200 mg QD (N=6) | Rucaparib 300 mg BID (N=5) | Rucaparib 300 mg QD (N=16) | Rucaparib 400 mg BID (N=2)
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib 200 mg BID (N=2) | Rucaparib 200 mg QD (N=6) | Rucaparib 300 mg BID (N=5) | Rucaparib 300 mg QD (N=16) | Rucaparib 400 mg BID (N=2)
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Aguesia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Breast atrophy (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 4 | 3 | 12 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 3 | 1
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Left chest wall tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Left rotator cuff tear (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 1 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Moist Desquamation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Olfactory nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 3 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Radiation skin reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Receding gum lower center jaw (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Seborrheic dermatitis (scalp) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Shingles (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 3 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT03542175/Prot_SAP_000.pdf